CLINICAL TRIAL: NCT06396819
Title: Topical Collagen-povidone Injection as an Alternative Treatment for Stenosing Tenosynovitis in Older Adults With Type 2 Diabetes Mellitus
Brief Title: Collagen-povidone for Diabetic Seniors' Tenosynovitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Collagen-Polyvidone-24
Record Dates: First submitted 2024-04-30; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Complications
Keywords: intervention; Stenosing Tenosynovitis; Collagen-Povidone
MeSH Terms: conditions — Diabetes Complications; Tendon Entrapment

STUDY DESIGN:
Intervention Model Description: A therapeutic intervention using povidone collagen vs. placebo was carried out, and the patients were recruited after meeting the inclusion criteria and divided into two randomized groups (Case vs Control). Application of collagen-povidone solution at a dose of 0.2 cc, compared with the application of physiological solution in the control group.
Who Masked: Participant
Masking Description: single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic intervention using povidone collagen (Experimental)
  Interventions: Drug: collagen-povidone solution
- Therapeutic intervention using placebo (Placebo Comparator)
  Interventions: Drug: collagen-povidone solution

INTERVENTIONS:
Drug: collagen-povidone solution — Application of collagen-povidone solution at a dose of 0.2 cc, compared with the application of physiological solution in the control group
  Other Names: Placebo

SUMMARY:
Diabetes affects 415 million adults globally, leading to hand issues. Povidone collagen shows promise in managing tenosynovitis. A clinical trial was conduced to compared its efficacy in adults over 60. It is shown that the intervention reduces pain, improves functionality, and grip strength with no complications. Collagen povidone holds potential for treating diabetic hand issues.

DETAILED DESCRIPTION:
A randomized clinical trial from January 2022 to January 2023 compared povidone collagen intervention with a placebo in adults aged 60 and above suffering from stenosing tenosynovitis. Participants were randomized into Case (collagen-povidone) and Control (physiological solution) groups. The study evaluated parameters like tenosynovitis, diabetes, pain, functionality, and grip strength.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of stenosing tenosynovitis
* Diagnostic of diabetes
* Adults aged 60 or older

Exclusion Criteria:

* Adults aged 60 or older

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Mean evolution time of tenosynovitis | 12 months
  Tenosynovitis should decreased its progression in the experimental group

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad de Investigación Biomédica 02, Unidad Médica de alta especialidad, Hospital de Especialidades Centro Médico Nacional de Occidente, Instituto Mexicano del Seguro Social, Guadalajara 44329, Mexico, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: Undecided